CLINICAL TRIAL: NCT03283891
Title: Effects on Nurses' Quality of Working Life and on Patients' Quality of Life of an Educational Intervention to Strengthen Humanistic Practice Among Haemodialysis Nurses in Switzerland: A Mixed Methods Cluster Randomised Controlled Trial
Brief Title: Effects on Nurses' Quality of Working Life of an Educational Intervention to Strengthen Their Humanistic Practice
Acronym: ExpCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Collaborators: Universite du Quebec en Outaouais (Other); Université de Sherbrooke (Other); School of Management and Engineering Vaud (Unknown); Université de Montréal (Other); University of Lausanne Hospitals (Other); Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Philippe Delmas, Inf, Ph.D, Ex.MBA., Professeur Ordinaire HES-SO, Institut et Haute Ecole de la Santé la Source
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FNS 10001C_172588
Record Dates: First submitted 2017-09-13; First posted 2017-09-14 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Patient-Centered Care
Keywords: Educational intervention; Watson's theory of human caring; Quality of working life of haemodialysis nurses; Quality of life of haemodialysis patients

STUDY DESIGN:
Intervention Model Description: Mixed methods cluster randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- educational intervention (Experimental): Various pedagogical activities to mobilise Watson's ten Carative Factors
  Interventions: Other: Educational intervention - humanistic nursing practice
- control (No Intervention): No intervention during the different times of measurement. Educational intervention will be delivered after the last measure.

INTERVENTIONS:
Other: Educational intervention - humanistic nursing practice — Four educational sessions:
  * Acquisition of core concepts of caring practice (I)
  * Acquisition of core concepts of caring practice (II)
  * Search for meaning: Influencing hope in persons through humanistic practice
  * Enacting different caring attitudes and behaviours in an intermediary simulation exercise with actor
  Arms: educational intervention

SUMMARY:
Haemodialysis (HD) patients constitute a vulnerable population with considerable health needs. They are often older persons with comorbid chronic conditions. Despite the substantial technical care they receive, these patients indicate that the quality of the human relationship that develops with nurses-the pivotal element in the care this population receives-can become therapeutic. This feature of the human relationship constitutes the cornerstone of the humanistic practice (caring practice) that all nurses should adhere to. However, according to some authors, such practice tends to fade over time. In 2012, a pilot study allowed to test an educational intervention based on Watson's Theory of Human Caring, the aim of which was to optimise nurses' humanistic practices. The intervention, first developed in Quebec and adapted in Switzerland by a committee of experts, was delivered to a group of nine HD nurses (Canton of Vaud, Switzerland) and evaluated. Preliminary results (qualitative and quantitative) showed the intervention to be highly feasible and acceptable. Moreover, in terms of preliminary outcomes, participating nurses appeared to strengthen their caring attitudes/behaviours toward HD patients post-intervention. Quantitative analyses of patients' questionnaires showed that HD patients perceived significant changes in nurses' caring attitudes/behaviours and maintained their level of quality of life (QoL) over time, which is a definite gain for this population. In light of these positive results, it is important to pursue this line of investigation in order to examine more accurately the intervention's effects on both nurses and patients. To this end, the investigators propose conducting a mixed-methods cluster randomised controlled trial (RCT) to assess the effects of an educational intervention to strengthen humanistic practice among nurses working in HD units in French Switzerland, on perceived quality of the nurse-patient relationship (NPR), nurses' team cohesion, nurses' quality of working life (QoWL), and HD patients' QoL. Knowledge acquired in the course of the study will contribute to strengthen nurses' humanistic practice, a key factor in HD patients' QoL.

ELIGIBILITY:
Inclusion Criteria:

* Nurses:

  1. have at least 6 months' work experience in the department;
  2. consent to take part in the study. In addition, nurses who intend to leave the HD unit in the 3 months to come will be excluded
* Patients

  1. be at least 18 years of age and under active treatment for at least 6 months;
  2. understand and read French;
  3. able to provide informed consent.

Exclusion Criteria:

* Nurses:

  1. intention to leave the HD unit in the 3 months after the beginning of the project
* Patients

  1. being diagnosed with dementia
  2. being a new HD patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Nurse-patient relationship (NPR) | 30 months
  NPR will be measured with the French version (EIIP-70) of the Caring Nurse-Patient Interaction Scale (CNPI-70). This tool comprises 70 items across 10 dimensions that capture each of Watson's 10 CF. It allows nurses to selfevaluate their frequency of caring attitudes/behaviours. More specifically, the EIIP-70 covers the following dimensions: humanism (6 items), hope (7 items), sensitivity (6 items), relationship (7 items), emotions (6 items), problem solving (6 items), teaching (11 items), assistance (10 items) and existential factors (6 items). Respondents must choose from five responses ranging from 1 (almost never) to 5 (almost always). This tool was validated on 377 nursing students and demonstrates good psychometric properties (Cronbach's alphas for the ten sub-dimensions range from .73 to .91).
Nurses' team cohesion | 30 months
  Team cohesion will be measured with the Group Environment Questionnaire (GEQ), which was subsequently adapted for work teams. Like the original, the French version contains 18 items and encompasses the four dimensions of team cohesion, namely, respondent's social-related attraction to the group (5 items, 1 of which is reverse scored), respondent's task-related attraction to the group (4 items, 2 of which are reverse scored), social-related group integration as perceived by respondent (4 items, 2 of which are reverse scored), and task-related group integration as perceived by respondent (5 items, 1 of which is reverse scored). The response scale ranges from 1 (strongly disagree) to 5 (strongly agree). The questionnaire was tested on a sample of nurses from another healthcare institution. No major comprehension difficulties emerged. Cronbach's alphas for the different dimensions run from 0.71 to 0.81.
Nurses' quality of working life (QoWL) - nurses | 30 months
  Quality of working life (QoWL) will be measured with a scale developed by Elizur and Shye (70), translated and validated in French. The scale is composed of 16 items exploring different dimensions of QoWL : psychological (items 1-4), physical (items 5-8), social (items 9-12) and cultural (items 13-16). Respondents must choose from six answers on a Likert scale ranging from "a very large part" to "very little".

SECONDARY OUTCOMES:
Hemodyalisis patients' quality of life (QoL) | 30 months
  Quality of life (QoL) of HD patients will be explored with a French version of the WHOQOL-BREF. This scale is a generic instrument that serves to explore perceived QoL and the impact of health problems on QoL. It comprises 26 items exploring four dimensions: physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items). It also contains two items measuring overall QoL, which is an added advantage of this instrument. Respondents must choose from five responses on a Likert scale ranging from 0 (not at all) to 5 (completely). The WHOQOLBREF yields an overall "QoL profile" score on a scale of 0 to 100, as well as scores for each dimension. A high score indicates a high perceived QoL. The French version translated and validated, and has shown perfectly satisfactory psychometric properties, and good acceptability by the population with a non-response rate below 5%.
Nurse-patient relationship (NPR) - patients | 30 months
  NPR will be explored with the French version (EIIP-70) (66) of the Caring Nurse-Patient Interaction Scale (CNPI-70) (for a description of dimensions, see Nurse section). Only the person addressed has been changed in order to adapt the items to the patient's viewpoint. The scale has been validated on a French population of patients living with HIV and presents perfectly satisfactory psychometric properties (Cronbach's alphas from 0.75 to 0.85). The scale allows HD patients to assess nurses' caring attitudes and behaviours.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Delmas, PhD, Principal Investigator — Haute Ecole de la Santé La Source
Locations (10):
- Switzerland (10):
  - Hôpital du Jura, Delémont, Canton of Jura
  - Centre hospitalier universitaire vaudois (CHUV), Lausanne, Canton of Vaud
  - Hôpital de Morges - Ensemble hospitalier de la Côte, Morges, Canton of Vaud
  - Hôpital intercantonal de la Broye (HIB), Payerne, Canton of Vaud
  - Établissements hospitaliers du Nord vaudois (eHnv), Yverdon-les-Bains, Canton of Vaud
  - Hôpital du Valais - Martigny, Martigny-Ville, Valais
  - Hôpital Riviera-Chablais (HRC), Monthey, Valais
  - Hôpital du Valais - Sierre, Sierre, Valais
  - Hôpital du Valais - Sion, Sion, Valais
  - Hôpitaux Universitaires de Genève (HUG), Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antonini M, Bellier-Teichmann T, O'reilly L, Cara C, Brousseau S, Weidmann J, Roulet-Schwab D, Ledoux I, Konishi M, Pasquier J, Delmas P. Effects of an educational intervention to strengthen humanistic practice on haemodialysis nurses' caring attitudes and behaviours and quality of working life: a cluster randomised controlled trial. BMC Nurs. 2021 Dec 20;20(1):255. doi: 10.1186/s12912-021-00729-6. PMID 34930206
- [Derived] Delmas P, O'Reilly L, Cara C, Brousseau S, Weidmann J, Roulet-Schwab D, Ledoux I, Pasquier J, Antonini M, Bellier-Teichmann T. Effects on nurses' quality of working life and on patients' quality of life of an educational intervention to strengthen humanistic practice among hemodialysis nurses in Switzerland: a protocol for a mixed-methods cluster randomized controlled trial. BMC Nurs. 2018 Nov 21;17:47. doi: 10.1186/s12912-018-0320-0. eCollection 2018. PMID 30479561